CLINICAL TRIAL: NCT06574685
Title: Efficacy of Twinkle Eyez Supplementation in Improving Ocular Health and Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ecolite Group (Industry)
Collaborators: UCSI University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ECO0001
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye Disease; Immunity
Keywords: Lutein; Zeaxanthin; Elderberry; Ocular Health; Immunity
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: One group intervention and one group placebo, consumption of supplements for 20 days.
Who Masked: Participant, Investigator
Masking Description: To maintain blinding, placebo supplements were identical in appearance to the intervention supplements, and investigators remained unaware of the participants' group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twinkle Eyez Supplementation (Experimental)
  Interventions: Dietary Supplement: Twinkle Eyez Supplementation
- Placebo control (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Twinkle Eyez Supplementation — The intervention supplement consisted of marigold extract, zeaxanthin, elderberry extract, bilberry extract, lycopene extract, multivitamin, silicon dioxide, inulin, and dextrose monohydrate, all in powder form and packaged in individual sachets (Twinkle Eyez™; Xmegami, Selangor, Malaysia). Each sachet contained 4.6 mg of lutein and zeaxanthin and 15.4 mg of elderberry extract.
  Arms: Twinkle Eyez Supplementation
Dietary Supplement: Placebo — The placebo supplement was identical in composition but excluded the active ingredients.
  Arms: Placebo control

SUMMARY:
This is a randomised, double-blind, placebo-controlled study that recruited 110 participants. The objectives of this study are to determine the dietary intake levels of lutein and zeaxanthin among precipitants. In additionally, this study also aimed to determine the efficacy of twinkle eyez supplementation in improving ocular health and immunity. The participant are required to take one sachet of twinkle eyez supplements or placebo for 20 days. The outcomes were assessed by food frequency questionnaire (FFQ), Ocular Surface Disease Index (OSDI), the Immune Status Questionnaire (ISQ), and the Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* presence of dry eye symptoms
* age 18 years or older
* ability to comprehend the study protocol and information provided by the investigators
* provision of informed consent.

Exclusion Criteria:

* ongoing medical treatment for ocular diseases or conditions
* use of certain medications, including hormone replacement therapy, antidepressants, and treatments for high blood pressure, acne, birth control, and Parkinson's disease
* history of eye surgery within the past three months
* pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Ocular Health | 20 days
  Ocular Surface Disease Index (OSDI) was used to assess the ocular health of participants. The OSDI, a validated 12-item questionnaire, assesses three subcategories: ocular symptoms, vision-related function, and environmental triggers. Each item is rated on a scale from 0 ('none of the time') to 4 ('all of the time'), with the final OSDI score calculated by summing the participant's responses
Ocular Health | 20 days
  Visual Analogue Scale (VAS) was used to assess the ocular health of participants. The VAS is a psychometric measuring instrument designed to document the characteristics of disease-related symptom severity or general wellbeing of an individual, often used in epidemiological and clinical research. Participants were asked to self-rate their current overall ocular health using a 10 cm VAS, where 0 indicated a very poor condition and 10 indicated an excellent condition.
Immunity | 20 days
  Immune Status Questionnaire (ISQ) and Visual Analogue Scale (VAS) was used to assess the immunity status of participants. The ISQ consists of seven items that assess the occurrence of various immune-related symptoms in the past. The total ISQ score was recoded onto a scale from 0 (very poor) to 10 (excellent).
Immunity | 20 days
  Visual Analogue Scale (VAS) was used to assess the immunity status of participants. The VAS is a psychometric measuring instrument designed to document the characteristics of disease-related symptom severity or general wellbeing of an individual, often used in epidemiological and clinical research. Participants were asked to self-rate their current overall immunity status using a 10 cm VAS, where 0 indicated a very poor condition and 10 indicated an excellent condition.

SECONDARY OUTCOMES:
Lutein and zeaxanthin intakes | 20 days
  Dietary intakes of lutein and zeaxanthin over the previous six months were assessed using a validated, simplified food frequency questionnaire (FFQ) tailored to include 30 food items known for their lutein and zeaxanthin content (1). For each food item, a specific serving size was provided, and participants reported their consumption frequency in terms of 'never' or the number of occasions per day, week, or month, as appropriate. The dietary intake of lutein and zeaxanthin was then calculated based on values from the United States Department of Agriculture-National Cancer Institute Carotenoids Database.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSI University, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request. All of the individual participant data collected during the trial, after deidentification will be shared upon reasonable request. Additional documents including study protocol, statistical analysis plan, informed consent form and clinical study report will also be made available. The data will be available immediately following publication with no end date. Data will be shared with anyone who wishes to access with reasonable request. The data can be used for any types of analyses.

REFERENCES:
- [Background] Cena H, Roggi C, Turconi G. Development and validation of a brief food frequency questionnaire for dietary lutein and zeaxanthin intake assessment in Italian women. Eur J Nutr. 2008 Feb;47(1):1-9. doi: 10.1007/s00394-007-0689-0. Epub 2007 Dec 28. PMID 18165856
- [Background] Miller KL, Walt JG, Mink DR, Satram-Hoang S, Wilson SE, Perry HD, Asbell PA, Pflugfelder SC. Minimal clinically important difference for the ocular surface disease index. Arch Ophthalmol. 2010 Jan;128(1):94-101. doi: 10.1001/archophthalmol.2009.356. PMID 20065224
- [Background] Verster JC, Kraneveld AD, Garssen J. The Assessment of Immune Fitness. J Clin Med. 2022 Dec 20;12(1):22. doi: 10.3390/jcm12010022. PMID 36614822
- [Background] Frings A, Ziaei M, Lundstrom M, Allan BD. The Vision Correction Questionnaire: an electronic patient-reported outcome measure for refractive surgery. J Cataract Refract Surg. 2022 Dec 1;48(12):1427-1432. doi: 10.1097/j.jcrs.0000000000001018. PMID 35858627